CLINICAL TRIAL: NCT05585502
Title: Impact of Muscle and Tendon Dysfunction on the Mechanics of Muscle Contraction and Locomotion Capacity in People With Type 2 Diabetes Mellitus, and Efficacy of a Passive Stretching Training Program to Counteract These Alterations
Brief Title: Impact of Muscle and Tendon Dysfunction in People With Type 2 Diabetes Mellitus
Acronym: T2D_MTU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universita di Verona (Other)
Collaborators: Azienda Ospedaliera Universitaria Integrata Verona (Other); University of Padova (Other)
Responsible Party: Principal Investigator, Paola Zamparo, Principal Investigator, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PZamparo
Record Dates: First submitted 2022-10-06; First posted 2022-10-18 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Muscle and tendon disorders; locomotion capacity; passive stretching
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Tendinopathy

STUDY DESIGN:
Intervention Model Description: The first part of the project is a cross-sectional design to test the association between: diabetic condition -> increase in muscle and tendon stiffness -> impairment of muscle-tendon function -> increase in the energy expenditure of locomotion (walking).
  The second part of the project is an intervention study that aims to test the effects of a stretching training program on muscle and tendon stiffness, muscle function and locomotor (walking) capacity.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): T2D patients and controls in the experimental group will undergo 50 telemedicine MOS sessions (15 minutes/day, 5 days/week, 10 weeks). Before the training period all subjects will participate to three different experimental sessions: during the first session a blood sample will be withdrawn and a skin biopsy will be taken; during the second session, muscle-tendon stiffness and muscle function will be evaluated; during the third session, the energy cost of walking will be determined at different speeds. After the training period and 5 weeks after the end of the training period, all subjects will repeat the second and the third sessions.
  Interventions: Other: Training (minute oscillation stretching)
- Control group (No Intervention): T2D patients and controls in the control group will not perform any specific training. However, they will participate to the same three sessions as the experimental group.

INTERVENTIONS:
Other: Training (minute oscillation stretching) — The training session involves the use of an elastic band that the subjects will use to induce passive ankle flexion /extensions (with a frequency of 1 Hz): 10 repetitions will be performed with 60 s exercise and 30 s of pause in-between. At the end of the session, the subjects will fill a diary with data of perceived intensity of exercise and localized ankle pain. The telemedicine session will be conducted by trained personnel.
  Other Names: Telemedicine training
  Arms: Training group

SUMMARY:
Diabetes is a chronic-degenerative metabolic disorder that has reached pandemic proportions mainly because of the increasing incidence and prevalence of type 2 diabetes mellitus (T2D).

Diabetes hurts cardiovascular function due to chronic hyperinsulinemia and hyperglycemia, along with increased advanced glycation end products (AGEs) causing nonenzymatic glycation of soft tissues, including muscle and tendon, and leading to an increase in muscle and tendon stiffness. In turn, the stiffening of the muscle-tendon complex reduces its capability to change in shape, affecting its potential for modulating the mechanical request during contraction (and locomotion), also increasing the metabolic demands during walking.

The present, multi-disciplinary, project combines several experimental methods and procedures to investigate the impact of muscle and tendon alterations on the mechanics of muscle contraction and locomotion capacity in T2D patients. In this project, we also propose a new training approach (minute oscillation stretching) to counteract these possible alterations (e.g. to decrease muscle and tendon stiffness).

DETAILED DESCRIPTION:
Diabetes is a chronic-degenerative metabolic disorder that has reached pandemic proportions, mainly because of the increasing incidence and prevalence of type 2 diabetes mellitus (T2D). According to the International Diabetes Federation (IDF, 2017), 425 million people suffer from diabetes worldwide and these may rise to 629 million in 2045 . Within this epidemiological perspective, diabetes emerges as one of the main metabolic disorders with substantial costs for regional and national sanitary systems.

Diabetes hurts cardiovascular function due to chronic hyperinsulinemia and hyperglycemia, along with increased advanced glycation end products (AGEs), pro-inflammatory cytokines, oxidative stress, obesity, dyslipidemia, and physical inactivity, all of which contribute to vascular dysfunction. In particular, several studies have shown that AGEs exert their negative effects through binding to a specific cellular receptor (RAGE), found in several cell systems such as monocytes and endothelial cells. However, little attention has been paid, so far, to alterations in the musculoskeletal system, which may contribute to the decline of the general state of health of diabetic people and may limit the therapeutic use of exercise in these subjects.

Diabetes causes non-enzymatic glycation of soft tissues, including muscle and tendon, leading to an increase in muscle and tendon stiffness. It was observed that Achilles tendon stiffness and skin connective tissue cross-linking are greater in diabetic patients compared to controls and it has been suggested that the elevated tendon stiffness may influence gait parameters. Indeed, during walking, diabetic patients display less Achilles tendon elongation, higher tendon stiffness and higher tendon hysteresis compared to healthy controls. The higher energy cost of walking in diabetic patients could thus be related to an impairment of the Achilles tendon function. The stiffening of the muscle, on the other hand, reduces its capability to change in shape, affecting its potential for modulating the mechanical request during contraction (and locomotion), also increasing the metabolic demands. Therefore, investigating the mechanical alterations caused by an increase in muscle and tendon stiffness could provide new insights into diabetes pathophysiology.

Training strategies able to reduce muscle and tendon stiffness are expected to improve muscle-tendon function and locomotor capability of diabetic patients. Even if strength and endurance training protocols allow to improve both blood glucose and muscle contractile function, they seem ineffective in reducing muscle and tendon stiffness in T2D patients. Notably, these training modalities present a significant dropout in the diabetic population, generally higher than 25%.

Static and dynamic stretching are effective in decreasing muscle and tendon stiffness but, in both cases, the decrease in stiffness is associated with a temporary decrease in muscle and tendon mechanical function.

Recently, a new stretching modality (minute oscillation stretching, MOS) was proposed that allows to condition the plantar-flexors muscle-tendon units by providing repetitive small longitudinal length changes using a passive stretch of the ankle joint. In young and healthy participants, a single session of unilateral MOS was sufficient to reduce muscle and tendon stiffness without affecting the muscle strength of the tested leg. Since the plantar-flexor muscles are the most important propulsive muscles for human locomotion, it can be expected that MOS training for the plantar-flexor may improve locomotor capability in diabetic people too. It is noteworthy that, due to the current SARS-Covid-19 pandemic, this training modality can be easily performed at home, under telemedicine training supervision, since no specific equipment is needed.

To summarize, a better understanding of the altered muscle and tendon mechanical properties in TD2 patients and of the effects that these alterations have on muscle contraction and locomotion capability can help in furthering our understanding on how diabetes affects physical activity, leading to inactivity. Finally, to investigate if and how these alterations could be reduced using a simple training program (MOS training), can help in designing more effective interventions, allowing to prescribe training modalities that these patients can easily perform (possibly limiting dropout).

ELIGIBILITY:
Inclusion Criteria:

* body mass index between 23 and 30 kg/m2
* moderate level of physical activity in the everyday life (assessed by means of the International Physical Activity Questionnaires, IPAQ)

Exclusion Criteria:

* neuropathy of nondiabetic origin
* severe neuropathy
* foot ulcers
* arterial insufficiency
* arthritis of the ankle/foot
* previous foot/knee surgery
* previous Achille tendon rupture
* previous Charcot foot
* cardiovascular and respiratory deficits that would impede the performance of the locomotion test
* insulin therapy

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-10 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Muscle and tendon stiffness differences between T2D patients and controls | Data will be collected at baseline (pre-intervention)
  Achilles tendon and muscle (gastrocnemius medialis) stiffness (units: Nm/mm) will be evaluated during isometric maximum voluntary contractions. Torque values (units: Nm) will be recorded using a dynamometer (Cybex Norm) whereas tendon elongation (units: mm) and muscle fascicle displacement (units: mm) will be recorded using an ultrasound scanner (MycrusExt, Telemed).

SECONDARY OUTCOMES:
Effect of training on muscle and tendon stiffness (in patients and controls) | Data will be collected at baseline, immediately after the intervention (10 weeks of training) and 5 weeks after the end of the intervention
  Achilles tendon and muscle (gastrocnemius medialis) stiffness (units: Nm/mm) will be calculated as described in outcome 1.
  Changes in these variables will be calculated between baseline and post training and between post training and washout.
Correlation between tissue glycation indicators (AGEs) and muscle-tendon stiffness in T2D patients and controls | Data will be collected at baseline (pre-intervention)
  AGEs (units: microgr/ml) will be assessed in blood samples and skin biopsies as a measure of long-term glycation.
  Achilles tendon and muscle (gastrocnemius medialis) stiffness (units: Nm/mm) will be calculated as described in outcome 1.
Correlation between tissue glycation indicators (RAGE) and muscle-tendon stiffness in T2D patients and controls | Data will be collected at baseline (pre-intervention)
  RAGE (units: picogr/ml) will be assessed in blood samples and skin biopsies as a measure of long-term glycation.
  Achilles tendon and muscle (gastrocnemius medialis) stiffness (units: Nm/mm) will be calculated as described in outcome 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Sezione di Scienze Motorie, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lapolla A, Traldi P, Fedele D. AGE in micro- and macroangiopathy. Contrib Nephrol. 2001;(131):10-21. doi: 10.1159/000060063. No abstract available. PMID 11125555
- [Background] Sell DR, Lapolla A, Odetti P, Fogarty J, Monnier VM. Pentosidine formation in skin correlates with severity of complications in individuals with long-standing IDDM. Diabetes. 1992 Oct;41(10):1286-92. doi: 10.2337/diab.41.10.1286. PMID 1397702
- [Background] Martinelli AR, Mantovani AM, Nozabieli AJ, Ferreira DM, Barela JA, Camargo MR, Fregonesi CE. Muscle strength and ankle mobility for the gait parameters in diabetic neuropathies. Foot (Edinb). 2013 Mar;23(1):17-21. doi: 10.1016/j.foot.2012.11.001. Epub 2012 Dec 27. PMID 23274122
- [Background] Couppe C, Svensson RB, Kongsgaard M, Kovanen V, Grosset JF, Snorgaard O, Bencke J, Larsen JO, Bandholm T, Christensen TM, Boesen A, Helmark IC, Aagaard P, Kjaer M, Magnusson SP. Human Achilles tendon glycation and function in diabetes. J Appl Physiol (1985). 2016 Jan 15;120(2):130-7. doi: 10.1152/japplphysiol.00547.2015. Epub 2015 Nov 5. PMID 26542519
- [Background] Petrovic M, Deschamps K, Verschueren SM, Bowling FL, Maganaris CN, Boulton AJM, Reeves ND. Altered leverage around the ankle in people with diabetes: A natural strategy to modify the muscular contribution during walking? Gait Posture. 2017 Sep;57:85-90. doi: 10.1016/j.gaitpost.2017.05.016. Epub 2017 May 19. PMID 28578139
- [Background] Petrovic M, Maganaris CN, Deschamps K, Verschueren SM, Bowling FL, Boulton AJM, Reeves ND. Altered Achilles tendon function during walking in people with diabetic neuropathy: implications for metabolic energy saving. J Appl Physiol (1985). 2018 May 1;124(5):1333-1340. doi: 10.1152/japplphysiol.00290.2017. Epub 2018 Feb 8. PMID 29420151
- [Background] Colberg SR, Sigal RJ, Fernhall B, Regensteiner JG, Blissmer BJ, Rubin RR, Chasan-Taber L, Albright AL, Braun B; American College of Sports Medicine; American Diabetes Association. Exercise and type 2 diabetes: the American College of Sports Medicine and the American Diabetes Association: joint position statement. Diabetes Care. 2010 Dec;33(12):e147-67. doi: 10.2337/dc10-9990. PMID 21115758
- [Background] Colberg SR. Key Points from the Updated Guidelines on Exercise and Diabetes. Front Endocrinol (Lausanne). 2017 Feb 20;8:33. doi: 10.3389/fendo.2017.00033. eCollection 2017. No abstract available. PMID 28265261
- [Background] Ikeda N, Inami T, Kawakami Y. Stretching Combined with Repetitive Small Length Changes of the Plantar Flexors Enhances Their Passive Extensibility while Not Compromising Strength. J Sports Sci Med. 2019 Feb 11;18(1):58-64. eCollection 2019 Mar. PMID 30787652
- [Background] Ikeda N, Yonezu T, Kawakami Y. Minute oscillation stretching: A novel modality for reducing musculo-tendinous stiffness and maintaining muscle strength. Scand J Med Sci Sports. 2021 Jan;31(1):104-114. doi: 10.1111/sms.13830. Epub 2020 Oct 7. PMID 32969540